CLINICAL TRIAL: NCT03382535
Title: The Well-being of Female Teacher's Voice During Teaching
Brief Title: Female Teacher's Voice During Teaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Tampere University (Other); Oulu University Hospital (Other); Umeå University (Other); Sonvox AB (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ooulu
Record Dates: First submitted 2017-12-01; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Functional Voice Disorder
Keywords: Voice disorder; Teacher's voice; Voice SPL (Voice sound pressure level); Voice F0 (Voice fundamental frequency); Voice therapy; Voice accumulator; Activity noise; Classroom
MeSH Terms: conditions — Voice Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants are randomly divided into three groups. Group 1: Voice therapy. Group 2: Voice therapy with carryover strategies (supplementary tasks and reminders).
  Group 3. Controls. No treatment during control period. After the control period participants are having Voice therapy or Voice therapy with carryover strategies.
Who Masked: Participant
Masking Description: Participants are not told what kind of a therapy they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Voice therapy (Active Comparator): An individually tailored voice therapy where the order and length of voice treatment methods will depend on the nature of each subject's voice problems. The intervention will take eight weeks and average of eight sessions (a' 45 min).
  Interventions: Behavioral: Voice therapy
- Voice therapy with carryover strategies (Experimental): A voice therapy as described above and an enhanced carryover program. By carryover we mean the process of extending new vocal skills outside the clinic. It includes supplementary tasks and reminders that will be tailored individually out of those direct and indirect methods that the subjects have adopted during therapy sessions. Additionally, the teachers will be doing vocal warm-up and relaxation exercises together with their pupils int the beginning and in the middle of a school day. The intervention will take eight weeks.
  Interventions: Behavioral: Voice therapy with carryover strategies
- Control group (Other): No intervention during eight weeks since this group will act as a temporary control group. After eight weeks, half of the participants in this group will be provided with Voice therapy and half with Voice therapy with carryover strategies.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Voice therapy — Voice therapy with direct and indirect therapy elements.
  Arms: Voice therapy
Behavioral: Voice therapy with carryover strategies — Voice therapy with direct and indirect therapy elements and supplementary tasks and reminders.
  Arms: Voice therapy with carryover strategies
Other: Control group — No therapy during eight weeks. After the control period half of the group will be provided with Voice therapy and half with Voice therapy with carryover strategies.
  Arms: Control group

SUMMARY:
Two voice therapy methods are compared. Activity noise levels and vocal load of teachers during teaching in primary school classrooms are evaluated. Acoustic and Workshop Interventions are implemented in order to reduce noise level during lesson.

DETAILED DESCRIPTION:
Due to the voice disorders, teachers are a major customer group for voice therapy. The main part of the study is comparison of two voice therapy methods.

There are several factors in the classroom that increase teacher's risk of voice disorders. One of the most significant is high noise level during lessons. This study explores the noise conditions the teachers are working in and how these conditions are related to the voice parameters and symptoms.

Finally, the study aims to determine whether classroom noise level can be lowered by improving classroom acoustics and by noise reducing workshops for teachers and pupils.

ELIGIBILITY:
Inclusion Criteria:

* Female teachers or teachers of special needs children from elementary schools
* Voice symptoms and willingness to participate in voice therapy
* Mother tongue Finnish
* No hearing loss, no need to use a hearing aid
* Non-smoking
* No neurological diseases
* No voice therapy during past year
* Successful phoniatric examination with rigid laryngoscopy or nasal endoscopy

Exclusion Criteria:

* Mother tongue other than Finnish
* Need to use a hearing aid
* Need for medical treatment in the larynx
* Abnormalities of the larynx
* Vocal cord paresis
* Laryngitis
* Posterior hypertrophy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-12-07 (Actual); Primary Completion 2014-12-20 (Actual); Study Completion 2016-06-14 (Actual)

PRIMARY OUTCOMES:
The change of the well-being of the teachers' voice. | Up to one week before the interventions, up to one week after the interventions, 6 months after the interventions, 1 year and 2 years after the interventions and up to one week after the control time (concerning control group).
  Subjective evaluation.Data collected with a questionnaire (Voice Activity and Participation Profile, VAPP) from the participants, answers given on a visual analogical scale (VAS) of 100 mm (0 = no disorder, 100 = extreme disorder).

CONTACTS AND LOCATIONS:
Overall Officials: Sirpa M Pirilä, MA, Study Chair — Ooulu